CLINICAL TRIAL: NCT03968874
Title: Improving Sleep, Sleep-related Outcomes, and Biomarkers in Veterans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miranda M Lim, Principal Investigator, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIRB #4268, eIRB #19411
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
Keywords: Veterans
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light box (Experimental): Commercially available lightbox emitting 10,000 lux of light. Subjects asked to use lightbox everyday for an hour for 4 weeks upon waking.
  Interventions: Device: Light box therapy
- Negative Ion Generator (Sham Comparator): Commercially available negative ion generator. Subjects asked to use everyday for an hour for 4 weeks upon waking.
  Interventions: Device: Negative Ion Generator

INTERVENTIONS:
Device: Light box therapy — The intervention is sitting in front of a lightbox for 1 hour in the morning upon waking up.
  Arms: Light box
Device: Negative Ion Generator — The intervention is sitting in front of a modified negative ion generator for 1 hour in the morning upon waking up.
  Arms: Negative Ion Generator

SUMMARY:
The primary purpose of this project is to determine the effect of morning bright light therapy (MBLT) on sleep in Veterans with traumatic brain injury (TBI). Secondarily, the project aims to identify blood-based brain biomarkers (BBBM) associated with sleep in Veterans.

Specific Aim 1. Determine the effect of MBLT on sleep quality in Veterans (primary outcome).

Specific Aim 2. Determine the effect of MBLT on downstream effectors of improved sleep, including cognition, mood, and quality of life measures in Veterans (exploratory outcomes).

Specific Aim 3. Determine the effect of MBLT on levels of specific BBBM related to sleep, and whether changes in specific BBBM predict response to MBLT (secondary outcome).

This study can now be completed 100% remotely.

DETAILED DESCRIPTION:
This project will utilize a biobehavioral intervention to improve sleep and apply a novel approach to measuring biomarkers in Veterans with TBI. The investigators will use morning bright light therapy (MBLT) to improve sleep. MBLT acts through intrinsically photosensitive retinal ganglion cells and has pleiotropic effects on sleep, circadian rhythms, cognition, mood, and pain through activation of brain circuits.

MBLT is a simple, cost-effective, home-based sleep intervention. It has been studied in a variety of neuropsychiatric populations, such as seasonal affective disorder, non-seasonal depression, Alzheimer's, Huntington's, Parkinson's disease, and schizophrenia. MBLT is an attractive intervention for TBI as patients typically report multiple concomitant symptoms including alterations in mood and alertness (daytime fatigue). One recent placebo-controlled study using MBLT reported improved fatigue in individuals with TBI. Moreover, MBLT has high patient acceptability and is scalable, owing to its ability to be rapidly implemented in any setting including in the home or in a rehabilitation facility.

To address the substantial limitation of using peripheral biomarkers to understand central pathophysiology in TBI, the investigators have developed a method to use blood-based brain biomarkers (BBBM) to track central pathophysiology and symptomatology of TBI and response to treatment. This method entails isolation of neuronally derived exosomes in peripheral blood. Exosomes are membrane bound structures that, instead of being delivered to lysosomes for destruction, reside in multivesicular bodies, fuse with the plasma membrane, and are exocytosed into extracellular spaces. Within the membrane of exosomes are various proteins present in the cell of origin; thus, the cargo of exosomes reflects the microenvironment from the site of exosome production. Exosomes hold promise in TBI since they can readily cross the blood brain barrier (BBB) and be isolated from peripheral circulation. Studying exosomes allows us to isolate those proteins that are routinely disrupted in patients with TBI and sleep disturbances, and to track changes in accordance with treatment condition over time.

In this project, the investigators will conduct a randomized controlled, single blinded trial in which Veterans with and without TBI will receive MBLT or modified negative ion generator; (see below for modification specifications) for 4-weeks. BBBM will be assessed in conjunction with MBLT/sham and neurobehavioral symptomatology. The investigators hypothesize that: 1) MBLT will be associated with improved sleep, and downstream effectors of improved sleep (i.e., cognition, mood, and quality of life), compared to the sham condition; 2) MBLT will show a correlation between BBBM and improved sleep, and levels of BBBM will predict those that respond to MBLT. This will provide novel insights into how these biomarkers relate to neuronal and behavioral changes following TBI and may inform trajectory of recovery.

The study can be completed 100% remotely, in person, or a combination of the two.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* English-speaking
* Accessible by phone

Exclusion Criteria:

* Decisional impairment
* Macular degeneration
* Bipolar disorder
* Shift work
* Currently using lightbox or negative ion generator

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline; after 4 weeks of intervention; and 2 months after the end of intervention
  Measures self-reported insomnia severity; total score range = 0-28 (higher total score = worse insomnia)

SECONDARY OUTCOMES:
Change in NFL, GFAP, UCH-L1, and total tau | Baseline; after 4 weeks of intervention; and 2 months after the end of intervention
  Change in neurofilament light chain (NFL), glial fibrillary acidic protein (GFAP), ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1), and total tau

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Lim, MD, PhD, Principal Investigator — Portland VA
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifiable data will be made available to qualified researchers on request to the study PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Information will be sent as soon as is practical and will be available as long as the PI is available.
Access Criteria: Legitimate research agenda, including but not limited to request to double-check presented or published results and novel analyses.